CLINICAL TRIAL: NCT03284983
Title: Split Scar Study to Assess Cosmetic Outcome From Differing Suture Spacing
Acronym: SFD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Silver Falls Dermatology (Other)
Collaborators: Samaritan Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB16-051
Record Dates: First submitted 2017-09-11; First posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Suture, Complication; Wound; Wound Complication; Wound Dehiscence; Wound of Skin; Surgery; Suture; Complications, Infection or Inflammation
MeSH Terms: conditions — Wounds and Injuries; Infections; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 10 mm suture spacing (Experimental): The investigators aim to determine how suture spacing affects cosmetic outcome of wound healing. One side (1/2 of the wound length) was sutured with 10 mm suture spacing
  Interventions: Other: Suture spacing for wound closure

INTERVENTIONS:
Other: Suture spacing for wound closure — The wound was divided in half and sutures were spaced 5mm or 10mm apart depending on side. The sutures were removed at 2-week follow-up appointment and photographs were taken. The Patient and Observer Scar Assessment Scale (POSAS) was then performed by both patient and physician.

SUMMARY:
The investigators wish to determine how suture spacing (5 mm vs. 10 mm) affects cosmetic outcome and development of "train tracking" in wounds. Linear wounds with sutures spaced closer together may not be as cosmetically appealing when compared to those that have larger spacing between sutures. Suturing closer together constricts blood flow and increases tension that ultimately results in more tissue necrosis and a less appealing outcome. The investigators also aim to conclude if 5 mm or 10 mm suture spacing results in less complications.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, at least 18 years of age, undergoing surgical excision of biopsy-proven skin cancers on the trunk or extremities at Silver Falls Dermatology & Allergy outpatient clinic in Salem, Oregon. Patients with elliptical excisions with length greater than 4.0 centimeters were included.

Exclusion Criteria:

* Patients with prior scars within 2.5cm of the proposed elliptical excision, failure to comply with wound care instructions or failure to follow up.

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-10-01 (Estimated); Study Completion 2017-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in cosmetic outcome of 5 mm versus 10 mm suture spacing on wound healing | 6 months
  The wound was divided in half by placing a single 4-0 Polysorb suture in the midpoint of the wound based on ruler measurement. Simple interrupted nylon sutures were spaced approximately 5mm or 10mm apart depending on side. The sutures were then removed at 2-week follow-up appointment. The Patient and Observer Scar Assessment Scale (POSAS) was then performed by both patient and physician. The observer scale consists of six items (vascularity, pigmentation, thickness, relief, pliability and surface area), and all items were scored on a scale from 1 ('like normal skin') to 10 ('worst scar imaginable'). The patient scale also includes six items (color, itch, pain, thickness, stiffness, and irregularity) and all items were scored on a similar scale from 1 ('like normal skin') to 10 ('worst scar imaginable').

SECONDARY OUTCOMES:
Change in wound complications of 5 mm versus 10 mm suture spacing on wound healing | 2 weeks
  Wounds were also assessed for complications. Difficulty removing sutures was assessed by presence of either one of the following: unable to directly visualize suture knot or need to probe into wound to remove suture. Wound dehiscence was defined as at least a 1mm separation of the wound edge for at least 50% of the length of the wound closure. Edge necrosis was defined as eschar and necrosis of the wound edge for at least 50% of the wound closure. Infection was defined as any wound that had redness, pain and exudate.

CONTACTS AND LOCATIONS:
Overall Officials: William Lear, MD, Principal Investigator — Silver Falls Dermatology
Locations (1):
- Silver Falls Dermatology, Salem, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dumville JC, Coulthard P, Worthington HV, Riley P, Patel N, Darcey J, Esposito M, van der Elst M, van Waes OJ. Tissue adhesives for closure of surgical incisions. Cochrane Database Syst Rev. 2014 Nov 28;2014(11):CD004287. doi: 10.1002/14651858.CD004287.pub4. PMID 25431843
- [Background] Bloemen MC, van Gerven MS, van der Wal MB, Verhaegen PD, Middelkoop E. An objective device for measuring surface roughness of skin and scars. J Am Acad Dermatol. 2011 Apr;64(4):706-15. doi: 10.1016/j.jaad.2010.03.006. Epub 2011 Jan 8. PMID 21216493
- [Background] Sagi HC, Papp S, Dipasquale T. The effect of suture pattern and tension on cutaneous blood flow as assessed by laser Doppler flowmetry in a pig model. J Orthop Trauma. 2008 Mar;22(3):171-5. doi: 10.1097/BOT.0b013e318169074c. PMID 18317050
- [Background] Braverman IM, Keh A, Goldminz D. Correlation of laser Doppler wave patterns with underlying microvascular anatomy. J Invest Dermatol. 1990 Sep;95(3):283-6. doi: 10.1111/1523-1747.ep12484917. PMID 2143522
- [Result] Shin TM, Bordeaux JS. How suture technique affects the cosmetic outcome of cutaneous repairs. J Drugs Dermatol. 2014 Aug;13(8):967-9. PMID 25116976